CLINICAL TRIAL: NCT01761695
Title: Prospective Observational Cohort Registry for Patients With Chronic Myeloid Leukemia at Asan Medical Center
Brief Title: Chronic Myelod Leukemia Registry at Asan Medical Center
Status: Terminated | Type: Observational
Why Stopped: The PI resigned the institute. The rest investigators at the institute decided to terminate the study.
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Dae-Young Kim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC-HEMREG-CML
Record Dates: First submitted 2013-01-03; First posted 2013-01-07 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Leukemia, Chronic Myeloid; Myeloid Leukemia, Chronic, Accelerated Phase; Myeloid Leukemia, Chronic, Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — Bone marrow aspirate or peripheral blood (for its mononuclear cells) will be collected, processed, and cryopreserved for future analysis of DNA or cell culture. Acquisition of biospecimens will be proceeded if patient agree with the informed consent for donation of biospecimen to 'Asan Medical Center Biomaterial Resource Banking Center'. This registry data will be used as a basic demographic and clinical information for the biospecimens.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- CML CP: Diagnosed as CML with chronic phase
  Interventions: Other: Diagnosed as CML
- CML AP: Diagnosed as CML with accelerated phase
  Interventions: Other: Diagnosed as CML
- CML BC: Diagnosed as CML with blast crisis
  Interventions: Other: Diagnosed as CML
- CML other: Diagnosed as CML, which is not included in any of other category
  Interventions: Other: Diagnosed as CML

INTERVENTIONS:
Other: Diagnosed as CML — All patients who will be enrolled in this prospective registry are confined to those who are diagnosed as chronic myeloid leukemia at Asan Medical Center, Seoul, Korea, from Jan 2013 till Dec 2047
  Other Names: Diagnosed as chronic myeloid leukemia

SUMMARY:
The investigators would like to propose a prospective longitudinal observational cohort study for patients who will be diagnosed and/or treated for chronic myeloid leukemia at Asan Medical Center, Seoul, Korea, to use the acquired data for fundamentals of other retrospective analysis.

DETAILED DESCRIPTION:
1. Acquisition of informed concent form
2. Data acquisition from medical record including

   * demographic / disease-associated factors
   * details of treatment, and its results
   * complications during treatment
   * genetic data
   * survival outcome (upto 30 years)
3. Accumulation of data for 30 years
4. Use of data for other retrospective analysis (including Asan Medical center Cell Banking basic data)

ELIGIBILITY:
Inclusion Criteria:

* All patients who are diagnosed and/or treated as chronic myeloid leukemia at Asan Medical Center
* 15 years of age and over
* All patients who give written consent according to guidelines at Asan Medical Center committee on human research

Exclusion Criteria:

* Patients who refuse to give consent to registering

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are diagnosed and/or treated with chronic myeloid leukemia at Asan Medical Center, Seoul, Korea
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Overall survival | 30 years

SECONDARY OUTCOMES:
Event-free survival | 30 years
  Definition of events will be as 'failure', 'progress to AP/BC', 'intolerant and medication change', and 'death from any cause'.
Failure-free survival | 30 years
  Failure will be defined as BCR-ABL elevation at 2 serial times, progression to AP/BC, loss of hematologic / cytogenetic response, any appearance of ABL kinase mutation, and clonal evolution.

CONTACTS AND LOCATIONS:
Overall Officials: Dae-Young Kim, MD, Principal Investigator — Assistant Professor
Locations (1):
- Asan Medical Center, Seoul, South Korea